CLINICAL TRIAL: NCT02038907
Title: A Phase II, Randomized, Controlled, Double-Blind, Dosage and Adjuvant Justification, Safety and Immunogenicity Trial of Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine Adjuvanted With or Without Monophosphoryl Lipid A and Aluminum Hydroxide in Adults
Brief Title: Safety and Immunogenicity of Norovirus GI.1/GII.4 Bivalent VLP Vaccine
Acronym: NOR-107
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-107; 2013-001419-64 (EudraCT Number); U1111-1147-3239 (Other: WHO)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers; Norovirus, Prevention
Keywords: Norovirus, vaccination
MeSH Terms: interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (14):
- GI.1/GII.4 (15/15) - MPL (50) (Experimental): Hepatitis A vaccine, intramuscular (IM), on Day 1, followed by norovirus bivalent virus like particle (VLP) vaccine (15 µg of GI.1 norovirus virus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 50 µg monophosphoryl lipid A (MLP) and 500 µg aluminum hydroxide, IM on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) - MPL (50) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MLP and 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (50/50) - MPL (50) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MLP and 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/15) - MPL (15) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) - MPL (15) (Experimental): IM hepatitis A vaccine on Day 1, followed by IM norovirus bivalent vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminum hydroxide, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (50/50) - MPL (15) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/15) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (50/50) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (50/150) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) - Al(OH)3 (167) (Experimental): Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminum hydroxide, IM, on Day 28.
  Interventions: Biological: Hepatitis A Vaccine; Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) x2 (Experimental): Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 1 and Day 28.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (50/150) x2 (Experimental): Norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, IM, on Day 1 and Day 28.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 (15/50) - Al(OH)3 (167) x2 (Experimental): Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminum hydroxide, IM, on Day 1 and Day 28.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine

INTERVENTIONS:
Biological: Hepatitis A Vaccine — Hepatitis A Vaccine IM injection
  Other Names: Havrix
  Arms: GI.1/GII.4 (15/15); GI.1/GII.4 (15/15) - MPL (15); GI.1/GII.4 (15/15) - MPL (50); GI.1/GII.4 (15/50); GI.1/GII.4 (15/50) - Al(OH)3 (167); GI.1/GII.4 (15/50) - MPL (15); GI.1/GII.4 (15/50) - MPL (50); GI.1/GII.4 (50/150); GI.1/GII.4 (50/50); GI.1/GII.4 (50/50) - MPL (15); GI.1/GII.4 (50/50) - MPL (50)
Biological: Norovirus Bivalent VLP Vaccine — Norovirus GI.1/GII.4 bivalent VLP vaccine IM injection

SUMMARY:
The purpose of this study is to select the optimal formulation of the norovirus vaccine from different concentrations of virus-like particles (VLP), Aluminum Hydroxide and MPL adjuvant (3-O-desacyl-4'-monophosphoryl lipid A) for further development.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine adjuvanted with aluminum hydroxide and with or without monophosphoryl lipid A (MPL). The norovirus vaccine is being tested to assess different formulations of the vaccine that will then be further developed.

This study will look at the number of antibodies to norovirus formed in people who take different formulations of the norovirus vaccine. The study will enroll approximately 420 patients. Participants will be randomly assigned (by chance) to one of fourteen treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need).

All participants will receive a vaccination on Day 1 and Day 28 of the study. Some treatment arms will receive one dose of the norovirus vaccine and some arms will receive two. In order to keep the treatment arms undisclosed to the patient and the doctor, those randomized to the one dose groups will receive a dose of Hepatitis A vaccine on Day 1 followed by the norovirus vaccine 28 days later. Participants will be asked to record any symptoms that may be related to the vaccine or the injection site in a diary card for 7 days after each vaccination.

This multi-centre trial will be conducted in Belgium. The overall time to participate in this study is up to 393 days. Participants will make 6 visits to the clinic, and will be contacted by telephone twice for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between 18 and 64 years of age at the time of enrollment.
2. In good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and clinical judgment of the investigator.
3. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Can comply with trial procedures and are available for the duration of the trial.

Exclusion Criteria:

1. Has received any vaccines containing Hepatitis A vaccine within the past 5 years.
2. Has contraindications, warnings, and/or precautions to vaccination with Havrix as specified within the Summary of Product Characteristics.
3. Has a clinically significant active infection (as assessed by the investigator) or oral body temperature 38°C (100.4°F) or higher within 3 days of the intended date of vaccination.
4. Has received antipyretic/analgesic medications within 24 hours prior to the intended vaccine administration.
5. Known hypersensitivity or allergy to investigational vaccine (including excipients of the investigational vaccine).
6. Has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.
7. Has a history of any progressive or severe neurologic disorder, seizure disorder, or Guillain-Barré syndrome.
8. Has history of any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
9. Known or inspected impairment/alteration of immune function, including the following:

   1. Chronic use of oral steroids (Equivalent to 20 mg/day prednisone for ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1.
   3. Receipt of immunostimulants within 60 days prior to Day 1.
   4. Receipt of parenteral, epidural, or intra-articular immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the trial.
   5. Receipt of immunosuppressive therapy within 6 months prior to Day 1.
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Heritable immunodeficiency.
10. Abnormalities of splenic or thymic function.
11. Has a known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
12. Has any serious chronic or progressive disease according to judgment of the investigator (eg, neoplasm, insulin dependent diabetes, cardiac, renal, or hepatic disease).
13. Has a body mass index (BMI) greater than or equal to 35 kg/m^2 (=weight in kg/[height in meters * height in meters]).
14. Is participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
15. Has received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine administration.
16. Is first degree relatives of individuals involved in trial conduct.
17. Has history of substance or alcohol abuse within the past 2 years.
18. If female, of childbearing potential, sexually active, and has not used any of the acceptable contraceptive methods for at least 2 months prior to trial entry.
19. Female participants of childbearing potential and sexually active, who refuse to use an acceptable contraceptive method from Day 1 through 6 months after the last dose of investigational vaccine.
20. Female participants who plan to donate ova from Day 1 through 6 months after the last dose of investigational vaccine.
21. Female participants with any positive pregnancy test.
22. Female participants who are pregnant or breastfeeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- Belgium (2):
  - Universiteit Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent

REFERENCES:
- [Derived] Leroux-Roels G, Cramer JP, Mendelman PM, Sherwood J, Clemens R, Aerssens A, De Coster I, Borkowski A, Baehner F, Van Damme P. Safety and Immunogenicity of Different Formulations of Norovirus Vaccine Candidate in Healthy Adults: A Randomized, Controlled, Double-Blind Clinical Trial. J Infect Dis. 2018 Jan 30;217(4):597-607. doi: 10.1093/infdis/jix572. PMID 29140444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Belgium from 28 March 2014 (first participants signed the informed consent form) to 19 June 2015.
Pre-assignment Details: Healthy volunteers were enrolled equally in 1 of 14 unique formulation treatment groups: 11 formulation arms received 1 dose and 3 formulation arms received 2 doses.
Period: Overall Study
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Started | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
Completed | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 27 | 28 | 29 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2 | Total
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31 | 420
Age, Continuous [Median (Full Range); unit: years] | 50.0 (14.70) [19 to 63] | 51.0 (14.36) [20 to 64] | 50.0 (12.95) [22 to 64] | 50.0 (14.95) [20 to 64] | 49.5 (13.79) [20 to 64] | 50.0 (14.39) [20 to 64] | 49.5 (14.19) [18 to 64] | 48.5 (14.13) [18 to 63] | 41.0 (14.82) [21 to 63] | 51.0 (15.26) [20 to 63] | 49.0 (15.41) [21 to 62] | 48.5 (14.05) [23 to 64] | 48.0 (15.06) [22 to 63] | 44.0 (16.11) [19 to 64] | 49.5 [18 to 64]
Age, Customized [Number; unit: participants]
  18-49 Years | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 16 | 15 | 15 | 15 | 14 | 15 | 16 | 210
  50-64 Years | 15 | 16 | 15 | 16 | 15 | 16 | 15 | 16 | 14 | 15 | 14 | 14 | 14 | 15 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 20 | 22 | 19 | 23 | 15 | 18 | 20 | 23 | 16 | 16 | 20 | 18 | 268
  Male | 12 | 10 | 10 | 9 | 11 | 8 | 15 | 14 | 9 | 7 | 13 | 12 | 9 | 13 | 152
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
  White | 29 | 30 | 30 | 30 | 30 | 29 | 30 | 32 | 28 | 29 | 29 | 28 | 29 | 31 | 414
Region of Enrollment [Number; unit: participants]
  Belgium | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31 | 420
Height [Median (Full Range); unit: cm] | 173.0 [156 to 187] | 167.0 [154 to 193] | 166.5 [153 to 191] | 167.0 [149 to 187] | 171.0 [155 to 186] | 169.0 [153 to 190] | 173.5 [154 to 189] | 169.5 [161 to 192] | 171.0 [153 to 193] | 167.0 [153 to 186] | 172.0 [156 to 199] | 171.5 [161 to 192] | 170.0 [153 to 187] | 175.0 [146 to 192] | 170.0 [146 to 199]
Weight [Median (Full Range); unit: kg] | 69.50 [49.4 to 105.2] | 65.60 [49.1 to 103.0] | 70.60 [50.8 to 104.0] | 66.60 [42.2 to 103.3] | 71.60 [47.6 to 101.9] | 68.50 [44.0 to 96.0] | 72.50 [45.8 to 104.5] | 74.35 [52.0 to 110.3] | 76.00 [54.8 to 101.2] | 69.85 [50.5 to 92.6] | 70.00 [49.6 to 94.0] | 75.50 [42.5 to 92.5] | 70.60 [49.2 to 111.8] | 69.90 [51.0 to 111.3] | 70.8 [42.2 to 111.8]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 25.22 [16.7 to 33.6] | 23.97 [18.9 to 34.2] | 26.11 [17.3 to 33.4] | 23.62 [18.7 to 33.7] | 24.51 [18.6 to 34.2] | 24.73 [17.6 to 34.4] | 24.40 [18.1 to 33.7] | 24.06 [17.8 to 33.2] | 26.06 [19.0 to 34.6] | 25.02 [20.0 to 34.4] | 23.66 [18.1 to 32.3] | 24.24 [14.9 to 32.7] | 23.19 [18.7 to 33.8] | 24.54 [17.9 to 33.5] | 24.52 [14.9 to 34.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Seroresponse (Pan-Ig ELISA)
Description: Seroresponse was defined as 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 56
Population: Full Analysis Set included all randomized participants who received at least one dose of trial vaccine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 31 | 30 | 31 | 30 | 32 | 28 | 30 | 26 | 28 | 29 | 30
percentage of participants | 43.3 [25.5 to 62.6] | 62.1 [42.3 to 79.3] | 46.4 [27.5 to 66.1] | 35.5 [19.2 to 54.6] | 80.0 [61.4 to 92.3] | 67.7 [48.6 to 83.3] | 30.0 [14.7 to 49.4] | 62.5 [43.7 to 78.9] | 42.9 [24.5 to 62.8] | 66.7 [47.2 to 82.7] | 46.2 [26.6 to 66.6] | 71.4 [51.3 to 86.8] | 69.0 [49.2 to 84.7] | 56.7 [37.4 to 74.5]

2. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site After Dose 1
Description: Solicited local AEs at injection site are defined as: pain, erythema, induration, and swelling that occurred within 7 days after each vaccination.
Time Frame: Days 1 through 7
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  Pain | 43.3 | 33.3 | 50.0 | 32.3 | 46.7 | 38.7 | 40.0 | 53.1 | 44.8 | 53.3 | 48.3 | 46.4 | 31.0 | 32.3
  Erythema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3.4 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site After Dose 2
Description: as for outcome 2
Time Frame: Days 28 through 34
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  Pain | 60.0 | 36.7 | 66.7 | 51.6 | 53.3 | 58.1 | 33.3 | 43.8 | 48.3 | 46.7 | 34.5 | 32.1 | 41.4 | 35.5
  Erythema | 0 | 0 | 3.3 | 0 | 0 | 0 | 0 | 0 | 3.4 | 3.3 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 3.3 | 0 | 6.7 | 0 | 0 | 0 | 3.4 | 3.3 | 0 | 0 | 0 | 0
  Swelling | 0 | 3.3 | 0 | 3.2 | 0 | 3.2 | 0 | 0 | 6.9 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) After Dose 1
Description: Solicited systemic AEs are defined as: headache, fatigue, myalgia, arthralgia, vomiting, and diarrhea that occurred within 7 days after each vaccination.
Time Frame: Days 1 through 7
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  Headache | 20.0 | 26.7 | 3.3 | 19.4 | 16.7 | 12.9 | 13.3 | 25.0 | 27.6 | 20.0 | 13.8 | 17.9 | 31.0 | 19.4
  Fatigue | 23.3 | 23.3 | 16.7 | 19.4 | 10.0 | 12.9 | 13.3 | 15.6 | 17.2 | 20.0 | 24.1 | 25.0 | 17.2 | 22.6
  Myalgia | 20.0 | 6.7 | 13.3 | 6.5 | 3.3 | 9.7 | 6.7 | 18.8 | 10.3 | 10.0 | 17.2 | 10.7 | 3.4 | 19.4
  Arthralgia | 0 | 3.3 | 6.7 | 0 | 3.3 | 0 | 3.3 | 6.3 | 6.9 | 3.3 | 3.4 | 3.6 | 3.4 | 3.2
  Vomiting | 0 | 3.3 | 0 | 0 | 0 | 3.2 | 0 | 0 | 0 | 3.3 | 3.4 | 0 | 0 | 0
  Diarrhea | 0 | 23.3 | 3.3 | 16.1 | 20.0 | 6.5 | 13.3 | 12.5 | 13.8 | 10.0 | 6.9 | 7.1 | 10.3 | 12.9

5. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) After Dose 2
Description: as for outcome 4
Time Frame: Days 28 through 34
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  Headache | 13.3 | 13.3 | 13.3 | 22.6 | 23.3 | 16.1 | 10.0 | 21.9 | 20.7 | 10.0 | 13.8 | 14.3 | 34.5 | 19.4
  Fatigue | 16.7 | 13.3 | 20.0 | 12.9 | 10.0 | 12.9 | 10.0 | 18.8 | 17.2 | 13.3 | 13.8 | 7.1 | 13.8 | 12.9
  Myalgia | 13.3 | 3.3 | 13.3 | 0 | 13.3 | 12.9 | 0 | 6.3 | 6.9 | 0 | 10.3 | 7.1 | 0 | 6.5
  Arthralgia | 0 | 3.3 | 3.3 | 0 | 3.3 | 3.2 | 0 | 3.1 | 0 | 3.3 | 3.4 | 3.6 | 0 | 3.2
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3.3 | 3.4 | 0 | 0 | 0
  Diarrhea | 3.3 | 10.0 | 16.7 | 12.9 | 16.7 | 9.7 | 6.7 | 15.6 | 17.2 | 10.0 | 3.4 | 7.1 | 6.9 | 3.2

6. Primary Outcome: Oral Body Temperature Within 7 Days After Dose 1
Description: Oral body temperature measurement is to be performed using the thermometer provided by the site for 7 days after each vaccination. The highest body temperature observed each day will be recorded on the Diary Card also provided by the site.
Time Frame: Days 1 through 7
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
degrees Celsius | 36.54 (0.294) | 36.76 (0.376) | 36.66 (0.345) | 36.71 (0.260) | 36.65 (0.388) | 36.67 (0.255) | 36.74 (0.323) | 36.63 (0.366) | 36.52 (0.405) | 36.77 (0.341) | 36.71 (0.404) | 36.61 (0.368) | 36.70 (0.362) | 36.61 (0.381)

7. Primary Outcome: Oral Body Temperature Within 7 Days After Dose 2
Description: as for outcome 6
Time Frame: Days 28 through 34
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 27 | 28 | 29 | 31
degrees Celsius | 36.54 (0.282) | 36.76 (0.301) | 36.68 (0.351) | 36.75 (0.466) | 36.60 (0.286) | 36.72 (0.317) | 36.71 (0.394) | 36.64 (0.342) | 36.59 (0.463) | 36.73 (0.293) | 36.68 (0.345) | 36.56 (0.351) | 36.76 (0.391) | 36.61 (0.386)

8. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study.
Time Frame: Day 1 up to Day 56
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants | 56.7 | 60.0 | 53.3 | 45.2 | 43.3 | 54.8 | 43.3 | 62.5 | 69.0 | 43.3 | 48.3 | 50.0 | 51.7 | 61.3

9. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Day 1 up to Day 393
Population: Safety population included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants | 6.7 | 0 | 16.7 | 6.5 | 3.3 | 0 | 10.0 | 9.4 | 3.4 | 3.3 | 3.4 | 7.1 | 3.4 | 3.2

10. Secondary Outcome: Percentage of Participants With a Seroresponse on Day 28, Day 208 and Day 393 (Pan-Ig ELISA)
Description: Seroresponse was defined as 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
  D=Day
Time Frame: Baseline and Days 28, 208 and 393
Population: Full Analysis Set included all randomized participants who received at least one dose of trial vaccine. "n" in the category is the number of participants with data available at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3] | 0 [0.0 to 11.6] | 0 [0.0 to 12.8] | 71.4 [51.3 to 86.8] | 79.3 [60.3 to 92.0] | 67.7 [48.6 to 83.3]
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,28) | 10.0 [2.1 to 26.5] | 17.2 [5.8 to 35.8] | 10.0 [2.1 to 26.5] | 19.4 [7.5 to 37.5] | 20.0 [7.7 to 38.6] | 20.0 [7.7 to 38.6] | 6.7 [0.8 to 22.1] | 34.4 [18.6 to 53.2] | 17.2 [5.8 to 35.8] | 23.3 [9.9 to 42.3] | 14.8 [4.2 to 33.7] | 32.1 [15.9 to 52.4] | 34.5 [17.9 to 54.3] | 35.7 [18.6 to 55.9]
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,29) | 17.2 [5.8 to 35.8] | 20.7 [8.0 to 39.7] | 13.3 [3.8 to 30.7] | 16.1 [5.5 to 33.7] | 10.0 [2.1 to 26.5] | 13.8 [3.9 to 31.7] | 10.3 [2.2 to 27.4] | 15.6 [5.3 to 32.8] | 6.9 [0.8 to 22.8] | 13.3 [3.8 to 30.7] | 7.4 [0.9 to 24.3] | 21.4 [8.3 to 41.0] | 20.7 [8.0 to 39.7] | 20.7 [8.0 to 39.7]

11. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in GI.1 VLP Antibody Titer (Pan-Ig ELISA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-like particle (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: Per-Protocol Set included all participants who received both doses of trial vaccine and who had no major protocol violations. "n" in the category is the number of participants with data available at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 12.8] | 6.9 [0.8 to 22.8] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.6] | 4.2 [0.1 to 21.1] | 85.7 [67.3 to 96.0] | 93.1 [77.2 to 99.2] | 93.3 [77.9 to 99.2]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 80.0 [61.4 to 92.3] | 89.7 [72.6 to 97.8] | 100.0 [87.7 to 100.0] | 89.7 [72.6 to 97.8] | 93.3 [77.9 to 99.2] | 96.8 [83.3 to 99.9] | 86.7 [69.3 to 96.2] | 87.5 [71.0 to 96.5] | 92.9 [76.5 to 99.1] | 90.0 [73.5 to 97.9] | 83.3 [62.6 to 95.3] | 85.7 [67.3 to 96.0] | 96.6 [82.2 to 99.9] | 86.7 [69.3 to 96.2]
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 60.0 [40.6 to 77.3] | 65.5 [45.7 to 82.1] | 67.9 [47.6 to 84.1] | 72.4 [52.8 to 87.3] | 70.0 [50.6 to 85.3] | 73.3 [54.1 to 87.7] | 66.7 [47.2 to 82.7] | 62.5 [43.7 to 78.9] | 85.7 [67.3 to 96.0] | 60.0 [40.6 to 77.3] | 54.2 [32.8 to 74.4] | 71.4 [51.3 to 86.8] | 75.9 [56.5 to 89.7] | 74.1 [53.7 to 88.9]
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 55.2 [35.7 to 73.6] | 46.4 [27.5 to 66.1] | 67.9 [47.6 to 84.1] | 69.0 [49.2 to 84.7] | 63.3 [43.9 to 80.1] | 65.5 [45.7 to 82.1] | 55.2 [35.7 to 73.6] | 53.1 [34.7 to 70.9] | 82.1 [63.1 to 93.9] | 43.3 [25.5 to 62.6] | 45.8 [25.6 to 67.2] | 64.3 [44.1 to 81.4] | 72.4 [52.8 to 87.3] | 78.6 [59.0 to 91.7]

12. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in GII.4 VLP Antibody Titer (Pan-Ig ELISA)
Description: The percentage of participants with a 4-fold rise or greater from in serum anti-norovirus antibody titers for GII.4 virus-like particle (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.9] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 3.1 [0.1 to 16.2] | 0 [0.0 to 12.8] | 3.3 [0.1 to 17.2] | 0 [0.0 to 14.2] | 78.6 [59.0 to 91.7] | 86.2 [68.3 to 96.1] | 70.0 [50.6 to 85.3]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 50.0 [31.3 to 68.7] | 65.5 [45.7 to 82.1] | 46.4 [27.5 to 66.1] | 41.4 [23.5 to 61.1] | 83.3 [65.3 to 94.4] | 71.0 [52.0 to 85.8] | 33.3 [17.3 to 52.8] | 71.9 [53.3 to 86.3] | 42.9 [24.5 to 62.8] | 73.3 [54.1 to 87.7] | 54.2 [32.8 to 74.4] | 78.6 [59.0 to 91.7] | 72.4 [52.8 to 87.3] | 63.3 [43.9 to 80.1]
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 16.7 [5.6 to 34.7] | 27.6 [12.7 to 47.2] | 7.1 [0.9 to 23.5] | 27.6 [12.7 to 47.2] | 36.7 [19.9 to 56.1] | 23.3 [9.9 to 42.3] | 16.7 [5.6 to 34.7] | 46.9 [29.1 to 65.3] | 14.3 [4.0 to 32.7] | 30.0 [14.7 to 49.4] | 16.7 [4.7 to 37.4] | 35.7 [18.6 to 55.9] | 41.4 [23.5 to 61.1] | 33.3 [16.5 to 54.0]
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 20.7 [8.0 to 39.7] | 32.1 [15.9 to 52.4] | 10.7 [2.3 to 28.2] | 27.6 [12.7 to 47.2] | 20.0 [7.7 to 38.6] | 17.2 [5.8 to 35.8] | 17.2 [5.8 to 35.8] | 21.9 [9.3 to 40.0] | 10.7 [2.3 to 28.2] | 13.3 [3.8 to 30.7] | 8.3 [1.0 to 27.0] | 28.6 [13.2 to 48.7] | 27.6 [12.7 to 47.2] | 21.4 [8.3 to 41.0]

13. Secondary Outcome: Geometric Mean Titer (GMT) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GI.1 VLP antibody titers as measured by pan-Ig ELISA.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 833.4 (4.64) | 790.3 (4.50) | 636.7 (4.60) | 647.6 (5.17) | 625.3 (2.96) | 520.3 (4.99) | 890.5 (4.75) | 842.9 (4.92) | 677.2 (3.75) | 827.3 (4.82) | 856.7 (5.34) | 741.5 (5.28) | 897.5 (3.74) | 742.7 (3.69)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 798.9 (4.66) | 737.9 (4.42) | 548.5 (4.47) | 806.6 (5.36) | 573.6 (3.08) | 514.6 (5.19) | 910.4 (4.37) | 821.5 (4.84) | 638.5 (3.90) | 780.6 (5.11) | 889.7 (5.34) | 14488.6 (3.00) | 20839.2 (1.96) | 15967.7 (2.39)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 14417.7 (2.74) | 14171.3 (2.76) | 17504.8 (2.64) | 14220.4 (3.23) | 13982.2 (2.33) | 18266.0 (1.99) | 16082.5 (2.07) | 15974.2 (3.95) | 25808.9 (2.55) | 15466.3 (2.59) | 14045.2 (2.94) | 12613.2 (2.46) | 17696.3 (1.92) | 12235.7 (2.11)
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,29) | 5725.2 (2.37) | 5069.7 (2.48) | 6084.3 (2.43) | 5613.9 (2.68) | 4467.6 (2.05) | 5106.4 (2.06) | 5660.5 (2.22) | 7174.8 (2.47) | 7542.0 (2.28) | 5361.1 (2.37) | 5162.8 (2.18) | 6863.9 (2.27) | 7459.1 (1.72) | 5912.6 (1.94)
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,29) | 3886.0 (2.98) | 3179.7 (2.78) | 4470.4 (2.55) | 5009.0 (2.80) | 3209.6 (2.54) | 3874.5 (2.55) | 4940.3 (2.48) | 4773.3 (2.62) | 5550.1 (2.70) | 3542.9 (2.54) | 3960.0 (2.55) | 4715.8 (2.51) | 5686.7 (2.17) | 4404.7 (2.19)

14. Secondary Outcome: Geometric Mean Titer (GMT) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GII.4 VLP antibody titers as measured by pan-Ig ELISA.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 1106.6 (4.68) | 1249.2 (3.45) | 1477.7 (4.13) | 1109.2 (4.10) | 921.7 (3.15) | 1130.9 (4.18) | 1340.4 (4.08) | 1238.6 (3.92) | 1201.2 (3.57) | 1473.2 (3.88) | 1832.3 (2.69) | 977.7 (3.73) | 1324.4 (3.34) | 1647.0 (3.39)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 1016.8 (5.56) | 1232.6 (3.46) | 1540.6 (3.83) | 1110.4 (3.84) | 839.4 (3.04) | 1097.8 (4.14) | 1268.1 (3.68) | 1311.0 (3.98) | 1139.9 (3.48) | 1494.7 (3.05) | 1924.8 (2.52) | 8459.4 (2.19) | 12901.7 (2.12) | 11116.3 (2.55)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 4595.7 (3.00) | 8636.7 (2.05) | 5750.4 (2.15) | 4391.5 (2.66) | 7545.2 (2.61) | 7802.7 (2.03) | 3444.6 (2.92) | 9945.7 (2.98) | 5129.9 (2.91) | 10624.2 (2.15) | 10034.2 (1.96) | 6622.0 (2.22) | 9995.5 (2.13) | 8164.0 (2.32)
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,29) | 2341.2 (3.93) | 3653.0 (2.24) | 2993.2 (3.61) | 2887.7 (2.78) | 2984.6 (2.62) | 3212.2 (2.44) | 2251.1 (3.15) | 5017.6 (2.82) | 2615.1 (2.91) | 4531.4 (2.21) | 4667.0 (2.20) | 3837.9 (2.30) | 4693.8 (2.52) | 4546.8 (2.26)
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,29) | 2236.5 (3.84) | 3103.0 (3.03) | 2450.2 (2.87) | 2175.3 (2.91) | 1946.4 (2.51) | 2173.7 (2.73) | 2267.2 (3.29) | 2969.9 (2.92) | 1898.2 (3.41) | 2550.0 (2.29) | 2871.1 (2.43) | 2425.1 (2.46) | 3133.0 (2.50) | 3060.7 (2.44)

15. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by pan-Ig ELISA.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
ratio
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 1.0 (1.13) | 0.9 (1.18) | 0.8 (1.50) | 1.2 (2.85) | 0.9 (1.26) | 1.0 (1.16) | 1.0 (1.36) | 1.0 (1.18) | 0.9 (1.28) | 0.9 (1.28) | 1.0 (1.58) | 19.5 (3.73) | 23.2 (3.00) | 22.0 (2.57)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 17.3 (3.69) | 18.8 (3.46) | 25.8 (3.09) | 22.4 (4.38) | 22.4 (3.02) | 35.1 (3.88) | 18.1 (4.35) | 19.0 (3.67) | 36.5 (4.85) | 18.7 (3.31) | 13.5 (3.07) | 17.0 (3.63) | 19.7 (2.78) | 16.8 (2.74)
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 6.9 (3.63) | 6.7 (3.71) | 9.3 (3.77) | 9.0 (4.32) | 7.1 (2.63) | 10.4 (3.79) | 6.4 (3.62) | 8.5 (3.90) | 10.7 (3.00) | 6.5 (2.96) | 5.2 (3.27) | 9.3 (3.57) | 8.3 (2.79) | 7.8 (3.52)
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 4.4 (3.27) | 4.1 (4.46) | 7.0 (3.56) | 8.0 (4.65) | 5.1 (2.41) | 7.4 (3.36) | 5.3 (3.40) | 5.7 (3.41) | 7.8 (2.87) | 4.3 (2.58) | 4.0 (3.08) | 6.4 (4.07) | 6.3 (2.95) | 6.1 (2.85)

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by pan-Ig ELISA.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
ratio
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0.9 (1.56) | 1.0 (1.14) | 1.0 (1.23) | 1.0 (1.21) | 0.9 (1.18) | 1.0 (1.13) | 0.9 (1.37) | 1.1 (1.57) | 1.0 (1.17) | 1.0 (1.58) | 1.0 (1.25) | 8.7 (3.25) | 9.7 (3.02) | 6.7 (3.11)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 4.2 (3.11) | 7.2 (2.98) | 4.0 (2.66) | 4.1 (2.97) | 8.2 (2.72) | 6.9 (3.31) | 2.6 (2.60) | 8.0 (3.36) | 4.0 (3.00) | 7.2 (3.38) | 4.7 (1.97) | 6.8 (2.99) | 7.5 (2.74) | 5.0 (2.70)
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 2.1 (2.45) | 3.0 (2.74) | 1.9 (1.96) | 2.6 (2.50) | 3.2 (2.36) | 2.7 (2.21) | 1.7 (2.17) | 4.1 (2.45) | 2.0 (2.06) | 3.1 (2.61) | 2.2 (1.92) | 3.9 (2.70) | 3.5 (2.24) | 2.5 (2.57)
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 1.9 (2.77) | 2.6 (3.20) | 1.7 (2.41) | 2.0 (2.33) | 2.1 (2.34) | 1.9 (1.99) | 1.6 (2.46) | 2.4 (2.40) | 1.5 (2.27) | 1.7 (2.41) | 1.4 (2.27) | 2.5 (2.60) | 2.4 (2.22) | 1.7 (2.64)

17. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GI.1 VLP and GII.4 VLP Antibody Titers (IgA ELISA)
Description: Percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 VLP and GII.4 VLP as measured by immunoglobulin A (IgA) enzyme-linked immunosorbent assay (ELISA) for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 3.03 [0.1 to 17.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3] | 0 [0.0 to 11.6] | 0 [0.0 to 12.8] | 71.4 [51.3 to 86.8] | 72.4 [52.8 to 87.3] | 64.5 [45.4 to 80.8]
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 53.3 [34.3 to 71.7] | 58.6 [38.9 to 76.5] | 39.3 [21.5 to 59.4] | 45.2 [27.3 to 64.0] | 70.0 [50.6 to 85.3] | 58.1 [39.1 to 75.5] | 36.7 [19.9 to 56.1] | 65.6 [46.8 to 81.4] | 42.9 [24.5 to 62.8] | 66.7 [47.2 to 82.7] | 50.0 [29.9 to 70.1] | 57.1 [37.2 to 75.5] | 51.7 [32.5 to 70.6] | 46.7 [28.3 to 65.7]
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 30.0 [14.7 to 49.4] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 25.0 [11.5 to 43.4] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 13.3 [3.8 to 30.7] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 6.5 [0.8 to 21.4] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected

18. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GI.1 VLP Antibody Titers (IgA ELISA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-like particle (VLP) as measured by immunoglobulin A (IgA) enzyme-linked immunosorbent assay (ELISA) for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 12.8] | 6.9 [0.8 to 22.8] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.6] | 4.2 [0.1 to 21.1] | 96.4 [81.7 to 99.9] | 100.0 [88.1 to 100.0] | 100.0 [88.4 to 100.0]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 93.3 [77.9 to 99.2] | 89.7 [72.6 to 97.8] | 100.0 [87.7 to 100.0] | 89.7 [72.6 to 97.8] | 96.7 [82.8 to 99.9] | 100.0 [88.8 to 100.0] | 90.0 [73.5 to 97.9] | 90.6 [75.0 to 98.0] | 96.4 [81.7 to 99.9] | 100.0 [88.4 to 100.0] | 87.5 [67.6 to 97.3] | 96.4 [81.7 to 99.9] | 100.0 [88.1 to 100.0] | 100.0 [88.4 to 100.0]
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 80.0 [61.4 to 92.3] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 71.9 [53.3 to 86.3] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 73.3 [54.1 to 87.7] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 54.8 [36.0 to 72.7] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected

19. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GII.4 VLP Antibody Titers (IgA ELISA)
Description: The percentage of participants with a 4-fold rise from or greater in serum anti-norovirus antibody titers for GII.4 virus-like particle (VLP) as measured by immunoglobulin A (IgA) enzyme-linked immunosorbent assay (ELISA) for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.7] | 0 [0.0 to 11.9] | 0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 3.1 [0.1 to 16.2] | 0 [0.0 to 12.8] | 3.3 [0.1 to 17.2] | 0 [0.0 to 14.2] | 75.0 [55.1 to 89.3] | 72.4 [52.8 to 87.3] | 63.3 [43.9 to 80.1]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 53.3 [34.3 to 71.7] | 65.5 [45.7 to 82.1] | 39.3 [21.5 to 59.4] | 51.7 [32.5 to 70.6] | 73.3 [54.1 to 87.7] | 58.1 [39.1 to 75.5] | 36.7 [19.9 to 56.1] | 68.8 [50.0 to 83.9] | 46.4 [27.5 to 66.1] | 66.7 [47.2 to 82.7] | 54.2 [32.8 to 74.4] | 60.7 [40.6 to 78.5] | 51.7 [32.5 to 70.6] | 46.7 [28.3 to 65.7]
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 36.7 [19.9 to 56.1] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 34.4 [18.6 to 53.2] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 23.3 [9.9 to 42.3] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | 16.1 [5.5 to 33.7] | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected | NA [NA to NA] — Data not collected

20. Secondary Outcome: Geometric Mean Titer (GMT) of GI.1 VLP Antibody Titers (IgA ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GI.1 VLP antibody titers as measured by IgA ELISA for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 52.9 (4.86) | 37.4 (3.59) | 42.1 (3.63) | 32.1 (5.26) | 30.1 (3.26) | 44.5 (6.06) | 53.6 (5.76) | 60.1 (6.45) | 36.8 (5.30) | 58.5 (4.08) | 47.0 (4.91) | 73.3 (5.24) | 40.8 (4.25) | 41.5 (3.74)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 48.9 (4.99) | 34.6 (3.38) | 41.2 (3.85) | 41.0 (4.38) | 29.4 (3.31) | 46.2 (6.22) | 54.4 (5.67) | 59.8 (6.23) | 37.8 (5.20) | 56.3 (3.95) | 57.0 (5.31) | 1649.9 (4.88) | 2148.2 (2.98) | 1703.2 (2.62)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30 | 1358.4 (4.02) | 996.2 (5.02) | 2223.3 (2.91) | 1068.7 (5.39) | 1368.6 (3.99) | 1849.8 (3.35) | 1594.9 (4.87) | 1435.5 (7.02) | 2074.3 (4.40) | 1510.6 (4.45) | 1131.2 (4.28) | 810.7 (5.58) | 922.6 (3.73) | 848.2 (3.63)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 302.5 (4.10) | NA (NA) — Data not collected | NA (NA) — Data not collected | 512.4 (5.85) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 224.0 (2.73) | NA (NA) — Data not collected | NA (NA) — Data not collected | 340.1 (3.91) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

21. Secondary Outcome: Geometric Mean Titer (GMT) of GII.4 VLP Antibody Titers (IgA ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GII.4 VLP antibody titers as measured by IgA ELISA for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 83.4 (6.63) | 113.6 (4.43) | 145.5 (4.72) | 119.5 (4.47) | 72.8 (4.64) | 114.6 (4.56) | 100.2 (4.47) | 133.0 (4.77) | 114.3 (4.65) | 158.5 (3.41) | 201.7 (3.30) | 105.9 (4.08) | 121.9 (4.16) | 174.5 (4.13)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 77.8 (6.49) | 110.0 (4.31) | 151.2 (4.70) | 125.3 (4.34) | 73.8 (4.42) | 116.3 (4.49) | 106.3 (4.05) | 139.2 (5.48) | 106.3 (4.71) | 164.8 (3.16) | 218.8 (3.07) | 953.5 (2.83) | 948.2 (2.52) | 1118.0 (2.91)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 495.7 (3.30) | 840.8 (2.87) | 583.7 (2.34) | 467.9 (2.79) | 803.3 (3.24) | 714.2 (2.44) | 336.7 (3.74) | 1088.9 (3.72) | 513.9 (3.82) | 1117.7 (3.03) | 1027.3 (2.36) | 578.8 (3.11) | 552.2 (2.60) | 691.2 (3.12)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 251.8 (3.94) | NA (NA) — Data not collected | NA (NA) — Data not collected | 427.9 (3.95) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 139.7 (4.07) | NA (NA) — Data not collected | NA (NA) — Data not collected | 273.4 (3.59) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

22. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (IgA ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by IgA ELISA for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
ratio
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0.9 (1.52) | 0.9 (1.49) | 1.0 (1.23) | 1.3 (2.65) | 1.0 (1.23) | 1.0 (1.14) | 1.0 (1.44) | 1.0 (1.10) | 1.0 (1.13) | 1.0 (1.46) | 1.2 (1.86) | 22.5 (2.95) | 52.7 (2.79) | 42.3 (2.39)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 25.7 (4.46) | 28.0 (4.40) | 49.2 (2.81) | 34.2 (5.55) | 45.4 (3.47) | 41.5 (3.50) | 29.8 (4.63) | 23.9 (4.13) | 52.1 (3.61) | 25.8 (3.15) | 20.8 (2.77) | 11.1 (2.19) | 22.6 (2.29) | 21.1 (2.81)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 10.0 (2.89) | NA (NA) — Data not collected | NA (NA) — Data not collected | 8.5 (3.77) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 7.4 (2.41) | NA (NA) — Data not collected | NA (NA) — Data not collected | 5.2 (3.34) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

23. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (IgA ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by IgA ELISA for all arms on day 28 and day 56 and for selected arms on day 208 and day 393.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
ratio
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0.9 (1.33) | 1.0 (1.42) | 1.0 (1.13) | 1.1 (1.27) | 1.0 (1.14) | 1.0 (1.09) | 1.1 (1.44) | 1.0 (1.60) | 1.0 (1.10) | 1.0 (1.36) | 1.0 (1.22) | 9.0 (2.85) | 7.8 (2.89) | 6.3 (3.11)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 5.9 (4.37) | 7.7 (3.92) | 3.6 (2.45) | 4.2 (2.54) | 11.0 (3.48) | 6.2 (3.36) | 3.4 (2.70) | 8.2 (3.36) | 4.0 (3.14) | 7.1 (2.81) | 4.9 (2.35) | 5.5 (4.74) | 4.5 (2.53) | 3.9 (2.41)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 3.5 (2.67) | NA (NA) — Data not collected | NA (NA) — Data not collected | 3.2 (2.44) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,31,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.9 (2.47) | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.9 (2.26) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

24. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Antibody Titers for GI.1 VLP and GII.4 VLP(HBGA)
Description: Percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 VLP and GII.4 VLP as measured by histoblood group antigen (HBGA) binding assay.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3] | 0 [0.0 to 11.6] | 0 [0.0 to 12.8] | 67.9 [47.6 to 84.1] | 62.1 [42.3 to 79.3] | 67.7 [48.6 to 83.3]
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 33.3 [17.3 to 52.8] | 55.2 [35.7 to 73.6] | 32.1 [15.9 to 52.4] | 35.5 [19.2 to 54.6] | 66.7 [47.2 to 82.7] | 51.6 [33.1 to 69.8] | 26.7 [12.3 to 45.9] | 59.4 [40.6 to 76.3] | 28.6 [13.2 to 48.7] | 60.0 [40.6 to 77.3] | 53.8 [33.4 to 73.4] | 75.0 [55.1 to 89.3] | 58.6 [38.9 to 76.5] | 56.7 [37.4 to 74.5]
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,28) | 10.0 [2.1 to 26.5] | 20.7 [8.0 to 39.7] | 16.7 [5.6 to 34.7] | 6.5 [0.8 to 21.4] | 13.3 [3.8 to 30.7] | 13.3 [3.8 to 30.7] | 20.0 [7.7 to 38.6] | 31.3 [16.1 to 50.0] | 20.7 [8.0 to 39.7] | 16.7 [5.6 to 34.7] | 7.4 [0.9 to 24.3] | 42.9 [24.5 to 62.8] | 34.5 [17.9 to 54.3] | 21.4 [8.3 to 41.0]
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,28) | 3.4 [0.1 to 17.8] | 13.8 [3.9 to 31.7] | 6.7 [0.8 to 22.1] | 3.2 [0.1 to 16.7] | 6.7 [0.8 to 22.1] | 3.4 [0.1 to 17.8] | 6.9 [0.8 to 22.8] | 9.4 [2.0 to 25.0] | 3.4 [0.1 to 17.8] | 3.3 [0.1 to 17.2] | 3.7 [0.1 to 19.0] | 7.1 [0.9 to 23.5] | 10.3 [2.2 to 27.4] | 7.1 [0.9 to 23.5]

25. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GI.1 VLP Antibody Titers (HBGA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-like particle (VLP) as measured by HBGA binding assay.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: Per-Protocol Set included all participants who received both doses of study drug and who had no major protocol violations. "n" in the category is the number of participants with data available at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0 [0.0 to 11.6] | 0 [0.0 to 11.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.9] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 12.8] | 0 [0.0 to 11.6] | 0 [0.0 to 14.2] | 82.1 [63.1 to 93.9] | 96.6 [82.2 to 99.9] | 93.3 [77.9 to 99.2]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 80.0 [61.4 to 92.3] | 79.3 [60.3 to 92.0] | 85.7 [67.3 to 96.0] | 82.8 [64.2 to 94.2] | 86.7 [69.3 to 96.2] | 87.1 [70.2 to 96.4] | 76.7 [57.7 to 90.1] | 78.1 [60.0 to 90.7] | 85.7 [67.3 to 96.0] | 90.0 [73.5 to 97.9] | 70.8 [48.9 to 87.4] | 100.0 [87.7 to 100.0] | 96.6 [82.2 to 99.9] | 93.3 [77.9 to 99.2]
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 53.3 [34.3 to 71.7] | 65.5 [45.7 to 82.1] | 67.9 [47.6 to 84.1] | 58.6 [38.9 to 76.5] | 43.3 [25.5 to 62.6] | 70.0 [50.6 to 85.3] | 60.0 [40.6 to 77.3] | 78.1 [60.0 to 90.7] | 82.1 [63.1 to 93.9] | 56.7 [37.4 to 74.5] | 33.3 [15.6 to 55.3] | 85.7 [67.3 to 96.0] | 93.1 [77.2 to 99.2] | 77.8 [57.7 to 91.4]
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 31.0 [15.3 to 50.8] | 32.1 [15.9 to 52.4] | 50.0 [30.6 to 69.4] | 37.9 [20.7 to 57.7] | 23.3 [9.9 to 42.3] | 37.9 [20.7 to 57.7] | 44.8 [26.4 to 64.3] | 53.1 [34.7 to 70.9] | 53.6 [33.9 to 72.5] | 26.7 [12.3 to 45.9] | 29.2 [12.6 to 51.1] | 50.0 [30.6 to 69.4] | 51.7 [32.5 to 70.6] | 46.4 [27.5 to 66.1]

26. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GII.4 VLP Antibody Titers (HBGA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GII.4 virus-like particle (VLP) as measured by HBGA binding assay.
  D=Day
Time Frame: Baseline and Days 28, 56, 208 and 393
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
percentage of participants
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 3.3 [0.1 to 17.2] | 0 [0.0 to 11.9] | 3.7 [0.1 to 19.0] | 0 [0.0 to 11.9] | 3.3 [0.1 to 17.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2] | 3.7 [0.1 to 19.0] | 3.3 [0.1 to 17.2] | 0 [0.0 to 14.2] | 82.1 [63.1 to 93.9] | 65.5 [45.7 to 82.1] | 70.0 [50.6 to 85.3]
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 46.7 [28.3 to 65.7] | 72.4 [52.8 to 87.3] | 39.3 [21.5 to 59.4] | 41.4 [23.5 to 61.1] | 80.0 [61.4 to 92.3] | 61.3 [42.2 to 78.2] | 26.7 [12.3 to 45.9] | 71.9 [53.3 to 86.3] | 35.7 [18.6 to 55.9] | 63.3 [43.9 to 80.1] | 66.7 [44.7 to 84.4] | 75.0 [55.1 to 89.3] | 58.6 [38.9 to 76.5] | 60.0 [40.6 to 77.3]
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 26.7 [12.3 to 45.9] | 31.0 [15.3 to 50.8] | 17.9 [6.1 to 36.9] | 20.7 [8.0 to 39.7] | 43.3 [25.5 to 62.6] | 20.0 [7.7 to 38.6] | 20.0 [7.7 to 38.6] | 43.8 [26.4 to 62.3] | 21.4 [8.3 to 41.0] | 33.3 [17.3 to 52.8] | 25.0 [9.8 to 46.7] | 50.0 [30.6 to 69.4] | 37.9 [20.7 to 57.7] | 22.2 [8.6 to 42.3]
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 13.8 [3.9 to 31.7] | 21.4 [8.3 to 41.0] | 3.6 [0.1 to 18.3] | 17.2 [5.8 to 35.8] | 23.3 [9.9 to 42.3] | 3.4 [0.1 to 17.8] | 10.3 [2.2 to 27.4] | 12.5 [3.5 to 29.0] | 10.7 [2.3 to 28.2] | 16.7 [5.6 to 34.7] | 4.2 [0.1 to 21.1] | 21.4 [8.3 to 41.0] | 24.1 [10.3 to 43.5] | 10.7 [2.3 to 28.2]

27. Secondary Outcome: Blocking Titers 50 (BT50) of Anti-Norovirus GI.1 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GI.1 VLP antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Baseline (Day 1) and Days 28, 56, 208 and 393
Population: Full Analysis Set included all participants who received at least one dose of trial vaccine. "n" in the category is the number of participants with data available at the given time-point.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 24.8 (2.75) | 18.7 (1.85) | 26.0 (2.73) | 26.8 (3.35) | 19.1 (1.68) | 24.8 (2.31) | 30.5 (3.04) | 24.5 (2.59) | 23.8 (2.46) | 23.2 (2.19) | 26.3 (2.68) | 23.1 (2.25) | 22.3 (2.26) | 20.6 (2.04)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 25.0 (2.60) | 18.6 (1.86) | 23.8 (2.44) | 26.7 (3.19) | 18.6 (1.70) | 23.0 (2.24) | 27.3 (2.46) | 25.1 (2.52) | 25.5 (2.52) | 24.8 (2.37) | 28.5 (2.66) | 347.6 (4.62) | 385.9 (3.64) | 391.1 (3.56)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 280.5 (3.94) | 236.3 (4.61) | 403.3 (3.74) | 286.9 (5.01) | 22.86 (3.94) | 356.4 (3.74) | 400.1 (3.33) | 412.9 (4.78) | 510.0 (4.36) | 247.2 (3.43) | 271.3 (5.00) | 398.6 (2.70) | 463.5 (2.32) | 355.8 (2.58)
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,29) | 130.0 (3.38) | 98.2 (3.46) | 159.0 (3.23) | 136.4 (3.67) | 80.1 (3.49) | 139.3 (2.68) | 159.8 (2.73) | 202.1 (3.34) | 208.6 (3.28) | 114.5 (2.89) | 107.9 (3.28) | 196.4 (2.86) | 219.2 (2.29) | 182.0 (2.40)
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,29) | 67.8 (3.78) | 51.3 (3.23) | 88.1 (3.54) | 74.8 (4.26) | 44.0 (3.39) | 71.9 (3.40) | 91.5 (3.14) | 107.5 (3.97) | 99.6 (4.09) | 55.0 (3.22) | 66.1 (3.86) | 103.4 (3.95) | 113.6 (3.30) | 81.0 (2.85)

28. Secondary Outcome: Blocking Titers 50 (BT50) of GII.4 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GII.4 VLP antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 27
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
titer
  D1 (n=30,30,30,31,30,31,30,32,29,30,29,28,29,31) | 66.0 (4.85) | 80.1 (3.44) | 115.3 (4.24) | 91.4 (4.15) | 60.9 (3.84) | 96.6 (4.03) | 80.7 (4.48) | 89.8 (4.41) | 96.2 (3.93) | 102.3 (3.39) | 121.9 (3.47) | 56.1 (3.48) | 92.0 (3.96) | 117.8 (3.91)
  D28 (n=30,30,29,31,30,31,30,32,28,30,27,28,29,31) | 69.3 (4.56) | 75.7 (3.63) | 124.9 (3.98) | 87.9 (3.75) | 67.7 (3.76) | 94.5 (4.30) | 74.6 (4.17) | 98.1 (5.11) | 92.9 (3.87) | 123.3 (3.25) | 117.6 (3.62) | 552.6 (3.65) | 688.4 (3.16) | 904.4 (2.67)
  D56 (n=30,29,28,31,30,31,30,32,28,30,26,28,29,30) | 336.9 (3.40) | 686.3 (3.47) | 429.0 (2.40) | 317.8 (2.94) | 675.7 (3.21) | 632.1 (2.11) | 189.2 (4.63) | 842.8 (3.23) | 360.1 (3.85) | 862.8 (3.12) | 778.0 (2.57) | 426.5 (3.46) | 596.3 (2.86) | 604.4 (2.91)
  D208 (n=30,29,30,31,30,30,30,32,29,30,27,28,29,29) | 186.7 (3.19) | 241.5 (3.24) | 244.6 (2.78) | 206.3 (2.84) | 229.9 (3.60) | 259.7 (2.66) | 142.5 (4.09) | 346.8 (2.92) | 201.0 (3.49) | 340.6 (2.60) | 324.6 (3.07) | 277.5 (2.53) | 350.9 (2.36) | 295.3 (3.07)
  D393 (n=29,29,30,31,30,29,29,32,29,30,27,28,29,28) | 120.5 (4.21) | 180.2 (3.95) | 123.5 (3.87) | 133.2 (3.81) | 104.7 (4.01) | 134.4 (3.74) | 109.3 (4.44) | 182.9 (3.60) | 121.9 (3.88) | 179.7 (2.53) | 209.0 (3.38) | 126.2 (3.56) | 171.2 (3.61) | 192.9 (3.52)

29. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (HBGA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 1.0 (1.30) | 1.0 (1.08) | 0.9 (1.30) | 1.0 (1.21) | 1.0 (1.37) | 0.9 (1.26) | 0.9 (1.59) | 1.0 (1.22) | 1.1 (1.37) | 1.1 (1.28) | 1.0 (1.31) | 15.0 (3.80) | 17.3 (3.02) | 19.3 (3.33)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 11.3 (4.25) | 13.2 (4.31) | 14.9 (3.54) | 10.0 (4.07) | 12.0 (3.36) | 14.3 (2.98) | 13.1 (3.96) | 16.9 (4.60) | 21.1 (3.72) | 10.7 (2.53) | 9.7 (4.29) | 17.2 (2.36) | 20.8 (2.20) | 17.9 (2.68)
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 5.2 (3.41) | 5.5 (3.18) | 6.0 (2.97) | 4.8 (2.91) | 4.2 (2.94) | 5.9 (2.00) | 5.2 (2.69) | 8.2 (3.14) | 8.6 (2.63) | 4.9 (2.24) | 3.7 (2.95) | 8.5 (2.52) | 9.8 (2.18) | 7.9 (2.21)
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 2.7 (3.29) | 2.7 (2.71) | 3.3 (2.87) | 2.6 (2.97) | 2.3 (2.65) | 3.0 (2.35) | 2.9 (2.61) | 4.4 (3.30) | 4.0 (3.10) | 2.4 (2.35) | 2.4 (2.73) | 4.5 (3.29) | 5.1 (2.81) | 3.8 (2.60)

30. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (HBGA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by the HBGA binding assay.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 1.1 (1.68) | 0.9 (1.59) | 1.0 (1.47) | 1.0 (1.73) | 1.1 (1.62) | 1.0 (1.38) | 0.9 (1.29) | 1.1 (1.89) | 1.0 (1.59) | 1.2 (2.45) | 1.0 (1.46) | 9.8 (3.48) | 7.5 (3.13) | 7.0 (2.96)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 5.1 (4.42) | 8.9 (3.31) | 3.6 (2.71) | 3.7 (3.43) | 11.1 (3.32) | 6.5 (3.33) | 2.3 (2.95) | 9.4 (3.95) | 3.5 (3.61) | 8.4 (3.59) | 6.0 (2.24) | 7.6 (3.19) | 6.5 (2.94) | 4.8 (2.46)
  D208 (n=30,29,28,29,30,30,30,32,28,30,24,28,29,27) | 2.8 (3.10) | 3.1 (2.51) | 2.0 (2.42) | 2.4 (2.58) | 3.8 (2.56) | 2.5 (1.99) | 1.8 (2.27) | 3.9 (3.03) | 2.0 (2.30) | 3.3 (2.66) | 2.5 (1.73) | 4.9 (2.72) | 3.8 (2.81) | 2.5 (2.35)
  D393 (n=29,28,28,29,30,29,29,32,28,30,24,28,29,28) | 1.7 (3.14) | 2.3 (2.42) | 1.0 (2.43) | 1.5 (2.56) | 1.7 (2.32) | 1.4 (1.82) | 1.3 (2.25) | 2.0 (2.59) | 1.3 (2.28) | 1.8 (2.11) | 1.6 (1.90) | 2.2 (2.70) | 1.9 (2.62) | 1.4 (2.23)

31. Secondary Outcome: GMFR of Antibody Titers of a Strain Not Represented in the Investigational Vaccine: GII.4 Cincinnati (HBGA)
Description: GMFR of anti-norovirus GII.4 Cincinnati antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 1.0 (1.17) | 1.0 (1.18) | 0.9 (1.12) | 1.0 (1.22) | 1.0 (1.11) | 0.9 (1.22) | 0.9 (1.18) | 1.0 (1.67) | 0.9 (1.98) | 1.0 (1.12) | 1.0 (1.13) | 7.4 (2.97) | 4.5 (2.94) | 5.7 (3.01)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 3.4 (2.91) | 5.1 (2.78) | 1.7 (1.81) | 2.6 (2.78) | 4.2 (3.20) | 3.7 (3.17) | 1.6 (2.06) | 5.9 (4.17) | 2.7 (3.16) | 4.6 (2.73) | 3.1 (2.36) | 4.6 (2.94) | 3.6 (2.62) | 4.0 (2.45)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.8 (2.34) | NA (NA) — Data not collected | NA (NA) — Data not collected | 2.4 (2.89) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.4 (2.08) | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.9 (2.56) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

32. Secondary Outcome: GMFR of Antibody Titers of a Strain Not Represented in the Investigational Vaccine: GII.4 Sydney (HBGA)
Description: GMFR of anti-norovirus GII.4 Sydney antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 0.9 (1.22) | 1.0 (1.26) | 0.9 (1.12) | 1.0 (1.18) | 0.9 (1.22) | 1.0 (1.09) | 0.9 (1.47) | 1.1 (1.91) | 1.0 (1.05) | 1.0 (1.25) | 1.0 (1.06) | 2.2 (2.48) | 2.5 (2.80) | 2.8 (2.77)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 1.5 (2.59) | 2.3 (2.10) | 1.3 (1.67) | 1.3 (1.48) | 2.0 (2.46) | 1.7 (1.82) | 1.1 (1.60) | 2.9 (3.50) | 1.6 (1.77) | 2.5 (2.62) | 2.0 (2.02) | 1.8 (2.25) | 1.9 (2.30) | 2.1 (2.25)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.4 (1.93) | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.6 (2.10) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.0 (1.78) | NA (NA) — Data not collected | NA (NA) — Data not collected | 1.4 (2.28) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

33. Secondary Outcome: GMFR of Antibody Titers of Strains Not Represented in the Investigational Vaccine: Cross-Protection Assays
Description: GMFR of anti-norovirus Cross-Protection Assays: GII.2 EC50, GI.3 EC50 and GII.4.2012 EC50 antibody titers as measured by HBGA binding assay. Data was collected for selected arms only.
  D=Day
Time Frame: Day 56
Population: Per-Protocol Set included all participants who received both doses of trial vaccine and who had no major protocol violations. Data was only collected for 2 of the arms.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (15/50)
Number analyzed (Participants) | 30 | 32
titer
  GII.2 EC50 | 1.1 (1.92) | 0.8 (3.73)
  GI.3 EC50 | 5.9 (3.23) | 3.0 (3.36)
  GII.4.2012 EC50 | 3.2 (2.50) | 4.1 (3.51)

34. Secondary Outcome: Blocking Titers 50 (BT50) of a Strain Not Represented in the Investigational Vaccine: GII.4 Cincinnati (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GII.4 Cincinnati antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D1 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 63.7 (4.34) | 75.1 (3.85) | 114.7 (4.28) | 85.8 (4.19) | 63.0 (4.08) | 89.1 (4.13) | 99.8 (4.47) | 85.0 (4.64) | 91.8 (4.02) | 112.6 (3.26) | 134.8 (3.07) | 54.0 (3.95) | 81.8 (3.86) | 93.2 (3.75)
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 63.6 (4.31) | 72.9 (3.95) | 113.8 (4.02) | 83.3 (4.05) | 61.7 (4.04) | 84.4 (4.23) | 90.5 (4.16) | 88.0 (5.49) | 78.6 (4.06) | 109.0 (3.25) | 130.6 (2.95) | 400.0 (3.57) | 366.9 (4.60) | 534.2 (3.17)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 217.3 (3.57) | 380.7 (3.61) | 200.3 (4.33) | 221.0 (3.66) | 263.7 (5.77) | 327.5 (4.12) | 161.5 (4.66) | 501.4 (5.07) | 248.5 (4.56) | 518.8 (3.40) | 415.5 (4.11) | 248.3 (4.01) | 296.5 (4.12) | 373.4 (3.40)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 113.5 (5.03) | NA (NA) — Data not collected | NA (NA) — Data not collected | 202.5 (4.06) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 88.9 (3.90) | NA (NA) — Data not collected | NA (NA) — Data not collected | 160.8 (3.96) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

35. Secondary Outcome: Blocking Titers 50 (BT50) of a Strain Not Represented in the Investigational Vaccine: GII.4 Sydney (HBGA)
Description: Blocking Titers 50 (BT50) of anti-norovirus GII.4 Sydney antibody titers as measured by HBGA binding assay.
  D=Day
Time Frame: Day 1 (Baseline) and Days 28, 56, 208 and 393
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 29 | 28 | 29 | 30 | 31 | 30 | 32 | 28 | 30 | 24 | 28 | 29 | 30
titer
  D1 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 35.0 (3.86) | 26.0 (2.30) | 43.3 (3.29) | 32.4 (3.24) | 28.3 (2.45) | 37.5 (3.18) | 29.7 (3.34) | 28.0 (2.93) | 32.2 (3.09) | 28.1 (2.31) | 32.3 (2.79) | 21.6 (2.11) | 29.7 (2.48) | 37.3 (3.42)
  D28 (n=30,29,27,29,30,31,30,32,27,30,24,28,29,30) | 32.6 (3.49) | 24.8 (2.29) | 42.5 (3.10) | 31.1 (3.12) | 26.4 (2.44) | 36.3 (3.09) | 25.9 (3.08) | 30.2 (3.87) | 32.9 (3.09) | 27.8 (2.28) | 31.8 (2.73) | 48.0 (3.37) | 75.1 (3.35) | 104.8 (3.35)
  D56 (n=30,29,28,29,30,31,30,32,28,30,24,28,29,30) | 53.5 (3.93) | 59.3 (2.79) | 56.7 (3.06) | 40.6 (3.37) | 55.5 (3.33) | 62.1 (3.26) | 31.2 (3.04) | 80.6 (4.37) | 51.2 (3.31) | 70.4 (3.22) | 64.4 (3.52) | 38.8 (2.98) | 56.7 (3.15) | 79.1 (3.18)
  D208 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 40.2 (3.14) | NA (NA) — Data not collected | NA (NA) — Data not collected | 44.2 (3.17) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected
  D393 (n=0,0,0,0,30,0,0,32,0,0,0,0,0,0) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | 28.5 (2.37) | NA (NA) — Data not collected | NA (NA) — Data not collected | 38.3 (2.87) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected

36. Secondary Outcome: Blocking Titers 50 (BT50) of a Strain Not Represented in the Investigational Vaccine: Cross-Protection Assay: GII.2 EC50 (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus Cross-Protection Assay: GII.2 EC50 antibody titers as measured by HBGA binding assay. Data was collected for selected arms only.
  D=Day
Time Frame: Day 1 (Baseline) and Day 56
Population: as for outcome 33
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (15/50)
Number analyzed (Participants) | 30 | 32
titer
  Day 1 | 266.2 (2.62) | 265.5 (4.79)
  Day 56 | 295.8 (2.31) | 216.5 (4.46)

37. Secondary Outcome: Blocking Titers 50 (BT50) of a Strain Not Represented in the Investigational Vaccine: Cross-Protection Assay: GI.3 EC50 (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus Cross-Protection Assay: GI.3 EC50 antibody titers as measured by HBGA binding assay. Data was collected for selected arms only.
  D=Day
Time Frame: Day 1 (Baseline) and Day 56
Population: as for outcome 33
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (15/50)
Number analyzed (Participants) | 30 | 32
titer
  Day 1 | 59.7 (2.98) | 74.1 (3.70)
  Day 56 | 350.5 (3.05) | 222.7 (5.09)

38. Secondary Outcome: Blocking Titers 50 (BT50) of a Strain Not Represented in the Investigational Vaccine: Cross-Protection Assay: GII.4.2012 EC50 (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus Cross-Protection Assay: GII.4.2012 EC50 antibody titers as measured by HBGA binding assay. Data was collected for selected arms only.
  D=Day
Time Frame: Day 1 (Baseline) and Day 56
Population: as for outcome 33
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (15/50)
Number analyzed (Participants) | 30 | 32
titer
  Day 1 | 45.5 (4.07) | 50.7 (5.10)
  Day 56 | 146.6 (3.11) | 208.5 (3.80)

39. Secondary Outcome: Percentage of Participants With Significant New Medical Conditions
Description: Significant new medical conditions will be evaluated by the investigator for the co-existence of any of the following conditions: Adverse events of special interest (AESIs) are predefined events for potential immune mediated disorders. All AESIs are medically evaluated to assess if they might indicate an immune-mediated disorder.
  Immune mediated events (IMEs) are AEs that represent a new diagnosis of a chronic medical condition that was not present or suspected prior to enrollment.
Time Frame: Day 1 up to Day 56
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants
  AESIs | 6.7 | 3.3 | 0 | 6.5 | 0 | 0 | 6.7 | 6.3 | 0 | 0 | 0 | 7.1 | 3.4 | 0
  IMEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Percentage of Participants With Any Adverse Event (AE) Leading to Withdrawal From the Study
Description: Withdrawal due to an AE will occur if the participant experiences an AE that requires early termination because continued participation imposes an unacceptable risk to the participant's health or the participants is unwilling to continue because of the AE.
Time Frame: Day 1 up to Day 56
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Number analyzed (Participants) | 30 | 30 | 30 | 31 | 30 | 31 | 30 | 32 | 29 | 30 | 29 | 28 | 29 | 31
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs 28 days after each vaccination (Day 1 to 56) and Serious Adverse Events (SAEs) throughout the trial (Up to Day 393)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | GI.1/GII.4 (15/15) - MPL (50) | GI.1/GII.4 (15/50) - MPL (50) | GI.1/GII.4 (50/50) - MPL (50) | GI.1/GII.4 (15/15) - MPL (15) | GI.1/GII.4 (15/50) - MPL (15) | GI.1/GII.4 (50/50) - MPL (15) | GI.1/GII.4 (15/15) | GI.1/GII.4 (15/50) | GI.1/GII.4 (50/50) | GI.1/GII.4 (50/150) | GI.1/GII.4 (15/50) - Al(OH)3 (167) | GI.1/GII.4 (15/50) x2 | GI.1/GII.4 (50/150) x2 | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/30 | 5/30 | 2/31 | 1/30 | 0/31 | 3/30 | 3/32 | 1/29 | 1/30 | 1/29 | 2/28 | 1/29 | 1/31
Other Adverse Events (participants affected / at risk) | 10/30 | 12/30 | 7/30 | 10/31 | 9/30 | 9/31 | 7/30 | 11/32 | 8/29 | 6/30 | 6/29 | 9/28 | 8/29 | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GI.1/GII.4 (15/15) - MPL (50) (N=30) | GI.1/GII.4 (15/50) - MPL (50) (N=30) | GI.1/GII.4 (50/50) - MPL (50) (N=30) | GI.1/GII.4 (15/15) - MPL (15) (N=31) | GI.1/GII.4 (15/50) - MPL (15) (N=30) | GI.1/GII.4 (50/50) - MPL (15) (N=31) | GI.1/GII.4 (15/15) (N=30) | GI.1/GII.4 (15/50) (N=32) | GI.1/GII.4 (50/50) (N=29) | GI.1/GII.4 (50/150) (N=30) | GI.1/GII.4 (15/50) - Al(OH)3 (167) (N=29) | GI.1/GII.4 (15/50) x2 (N=28) | GI.1/GII.4 (50/150) x2 (N=29) | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2 (N=31)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GI.1/GII.4 (15/15) - MPL (50) (N=30) | GI.1/GII.4 (15/50) - MPL (50) (N=30) | GI.1/GII.4 (50/50) - MPL (50) (N=30) | GI.1/GII.4 (15/15) - MPL (15) (N=31) | GI.1/GII.4 (15/50) - MPL (15) (N=30) | GI.1/GII.4 (50/50) - MPL (15) (N=31) | GI.1/GII.4 (15/15) (N=30) | GI.1/GII.4 (15/50) (N=32) | GI.1/GII.4 (50/50) (N=29) | GI.1/GII.4 (50/150) (N=30) | GI.1/GII.4 (15/50) - Al(OH)3 (167) (N=29) | GI.1/GII.4 (15/50) x2 (N=28) | GI.1/GII.4 (50/150) x2 (N=29) | GI.1/GII.4 (15/50) - Al(OH)3 (167) x2 (N=31)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 2 | 1 | 4 | 2 | 1 | 0 | 0 | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 2 | 2 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2
Headache (Nervous system disorders) | 3 | 8 | 3 | 3 | 3 | 3 | 0 | 0 | 1 | 1 | 4 | 2 | 2 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2 | 3 | 1 | 1 | 3 | 0 | 1 | 3 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.